CLINICAL TRIAL: NCT01385943
Title: VivaNet Study. A Multicenter Study of Confocal Reflectance Microscopy in Telemedicine
Acronym: EUNET
Status: Withdrawn | Type: Observational
Why Stopped: Study not launched due to logistical issues that could not be resolved.
Sponsor: Lucid, Inc. (Industry)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital Universitario Ramon y Cajal (Other); Hospital del Mar (Other); University of Modena and Reggio Emilia (Other); Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Organization: Lucid (Unknown)
Other Study IDs: 2009/4714
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Skin Cancer; Skin Lesions
Keywords: Reflectance Confocal Microscopy; Dermoscopy; Clinical Photos; Telemedicine
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Cutaneous tissue specimens in the form of histopathology slides and tissue blocks, clinical pictures, dermoscopic pictures and confocal microscopy images
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Skin Cancer: Patients from dermatology practices throughout Europe that have a skin lesion or tumor requiring a biopsy for diagnosis.

SUMMARY:
The goal of this study is to test a protocol that uses clinical pictures, confocal reflectance microscopy images and dermoscopic information in a telemedicine platform. This protocol will test the technologies and diagnostic performance of dermoscopy and confocal reflectance microscopy in a randomized prospective multicenter study in five different centers in Europe.

DETAILED DESCRIPTION:
In vivo confocal reflectance microscopy (CRM) is a non-invasive method for the in vivo (without cutting into the skik) examination of skin tumors. CRM produces cellular images with resolution comparable to histopathology. The procedure is painless, takes about ten minutes and has no documented side effects. Studies performed in the past decade have correlated CRM features in benign (non-cancerous) and malignant (cancerous) skin lesions such as moles and melanomas, as well as features of inflammatory lesions (such as allergic skin reactions) to histopathology.

Dermoscopy is a complementary technique that has been proven to be superior to the naked eye for the diagnosis of melanoma as well as some non-melanocytic skin tumors. Recently, correlation of dermoscopic and CRM structures has focused interest in the research in different groups that show that both are complementary and render in combination a better understanding of skin disease.

In this study, patients from several research centers in Europe, with lesions suspicious for malignancy and scheduled for biopsy will be asked if they would like to participate in the study. If they consent to the study, first, a clinical photograph will be taken of the lesion. Second, a dermoscopic image will be taken of the lesion, and third, CRM images will be taken of the lesion. Finally, the biopsy will be performed as per the standard of care. The images will be sent over a secure, private internet connection to physicians specially trained in the interpretation of dermoscopic and CRM images. An electronic report will be completed and returned to the Study Coordinator, who will correlate the results with the histopathologic diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Any skin tumor considered suspicious for malignancy under clinical non-aided examination
* Histopathologic study of the tumor or short term follow up (3 months) to confirm benignity
* Clinical information and images available
* Adequate imaging by dermoscopy and CRM according to the protocol of the study
* Consent form signed by the patient

Exclusion Criteria:

* Lesions with ulcerations obscuring more than 75% of the confocal mosaic field of view.
* Lesions with clinically appreciable scar.
* Lesions in locations not amenable to imaging with the confocal microscope.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients from private dermatology clinics and university dermatology practices throughout Europe that have a skin lesion suspicious for malignancy under clinical non-aided examination.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy, in terms of sensitivity, specificity, positive and negative predictive values with respect to histopathologic diagnosis. | Study participation will be no longer than three months for patients requiring follow up, and no longer than one office visit (approximately one hour) for patients being biopsied the same day they are imaged.
  Clinical pictures, dermoscopic pictures, confocal images and tissue biopsy will be obtained in a single study visit unless the physician determines that short-term (3 months) follow up is more appropriate, then the patient will be asked to return in three months for additional examination.

SECONDARY OUTCOMES:
Differences between dermoscopy/confocal microscopy, and dermoscopy plus confocal microscopy | Study participation will be no longer than three months for patients requiring follow up, and no longer than one office visit (approximately one hour) for patients being biopsied the same day they are imaged.
  Clinical pictures, dermoscopic pictures, confocal images and tissue biopsy will be obtained in a single study visit as described under Primary Outcomes, unless the physician determines that short-term (3 months) follow up is more appropriate, then the patient will be asked to return in three months for additional examination.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Malvehy, MD, Principal Investigator — Hospital Clinic of Barcelona, Spain; Giovanni Pellacani, MD, Principal Investigator — Policlinico Hospitale in Modena, Italy
Locations (6):
- Italy (2):
  - University of Modena and Reggio Emilia, Modena
  - Arcispedale Santa Maria Nuova, Reggio Emilia
- Spain (4):
  - Department of Dermatology, Hospital del Mar, Barcelona
  - Diagnosis Dermatologica, Barcelona
  - Hospital Clinic of Barcelona, Barcelona
  - Hospital Ramón y Cajal, Madrid